CLINICAL TRIAL: NCT02319876
Title: Expression and the Clinical Significance of TIM-3 on Lymphocytes During Sepsis
Brief Title: Expression of TIM-3 on Lymphocytes in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiaoming Deng, professor and chief, Changhai Hospital
Other Study IDs: TIM3-SEPSIS; 81201492 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-06

CONDITIONS: Sepsis; Immunosuppression
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample was collected to examine TIM-3 on CD4+ and CD8+ lymphocytes, and CD14+ monocytes. Monocyte HLA-DR will also be determined.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Severe sepsis: Patients with severe sepsis
- SIRS patient: Patients after elective surgeries presented with SIRS but without sepsis
- Volunteer: Volunteers

SUMMARY:
The current project was designed to examine the express TIM-3 on lymphocytes and monocytes and its role in immunosuppression during sepsis.

DETAILED DESCRIPTION:
Immunosuppression is the leading cause of death in septic patients.Lymphocyte apoptosis has been recognized as an important step in the pathogenesis of sepsis. Previous studies indicated that T cell immunoglobulin and mucin protein 3 (TIM-3) is a type I cell surface protein and was identified as a marker of lymphocyte dysfunction. The current project was designed to examine the express TIM-3 on lymphocytes and monocytes and its further role in immunosuppression during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe sepsis
* patients undergo invasive spine surgery
* healthy volunteers

Exclusion Criteria:

* patients with immunodeficient diseases
* patients who accept glucocorticoid or immunosuppressant
* patients with an age older than 18 years
* patients providing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU at Changhai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
TIM-3 expression on CD4+, CD8+ T cells and CD14+ monocytes | within 24h after recruitment
  TIM-3 level on T cells was compared between different populations.

SECONDARY OUTCOMES:
28-day mortality | 28 days after diagnosis of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Deng, M.D., Ph.D., Principal Investigator — Changhai Hospital
Locations (1):
- Anesthesiology and Intensive Care, Changhai Hospital, Shanghai, Shanghai Municipality, China